CLINICAL TRIAL: NCT04218331
Title: Predicting & Optimizing Language Outcomes in Minimally Verbal Children With Autism Spectrum Disorder: Boosting Language Outcomes of Minimally Verbal Children With ASD
Brief Title: Boosting Language Outcomes of Minimally Verbal Children With ASD (BLOOM)
Acronym: BLOOM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor/PhD, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-000806
Record Dates: First submitted 2019-11-19; First posted 2020-01-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: PROMPT; JASPER; speech; autism; ELSA-T
MeSH Terms: conditions — Autism Spectrum Disorder; Speech; Autistic Disorder | interventions — Activator Appliances

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JASPER only (Experimental): This group will consist of the child and therapist having one-on-one, JASPER sessions, twice a week.
  Interventions: Behavioral: JASPER
- JASPER + PROMPT (Active Comparator): This group will consist of the child and therapist having one-on-one, JASPER sessions plus Prompts for Restructuring Oral Muscular Phonetic Targets (PROMPT), twice a week.
  Interventions: Behavioral: JASPER; Behavioral: PROMPT

INTERVENTIONS:
Behavioral: JASPER — JASPER is a developmentally anchored behavioral intervention that assumes that communication develops from social interactions in which specific social engagement strategies, symbolic representations, and early communication forms are modeled and naturally reinforced by the adult's responses to the child. The adult referred in this condition is the clinician/therapist.
Behavioral: PROMPT — PROMPT is a multidimensional oral-motor approach to speech production disorders.
  Arms: JASPER + PROMPT

SUMMARY:
In this project, the investigator will test the effect of augmenting an evidence based joint attention intervention (JASPER) with a motor-sound system intervention (PROMPT) compared to JASPER only on speech and language outcomes. The investigator will model change over a year to determine the percentage of children who cross the hurdle from single words to word combinations by Kindergarten. The proposed research will foster the understanding of the mechanisms underlying speech heterogeneity in ASD, thereby ultimately contributing to the development of more personalized, efficacious interventions.

Upon qualification to the study (after entry assessments), the child will be randomized to receive JASPER alone (play-based intervention) or JASPER plus PROMPT (both play-based and speech-based interventions). The active intervention will last for 12 weeks, 60 minute sessions twice a week. There are assessments scheduled at entry (6.5 hours), end of study (exit-2.5 hours), 3 month follow up (2 hours), and when the child turns 6 years of age (2 hours). The total time commitment per participant is 37 hours.

DETAILED DESCRIPTION:
Children will be recruited through local school districts and early intervention service providers, approximately 20 children per year for a total of 80 children. Parents interested in the study will call the lab and be screened. If children pass the screen, they will be invited to go to UCLA for a series of assessments. The process will take 2-3 days. The following assessments and data will be collected: ADOS-2, ADI-R, Mullen Scales of Early Learning (MSEL), Demographic & Medical Questionnaires, Vineland-III Interview, ELSA Language Sample, PLS-5,SPA, Repetitive Behaviors RBS-R, SSP, ABC-2, ESCS, BOSCC, KSPT, EEG, and saliva sample. Eligibility for the study will then evaluated. Each child's clinical diagnosis of ASD will be validated by administration of the Autism Diagnostic Observation Schedule-2 (ADOS-2) and the Autism Diagnostic Interview-Revised (ADI-R) by a research-reliable lab staff. Children will participate in a language sample (eligible if < 20 words), and the Mullen Scales of Early Learning (MSEL) to evaluate nonverbal mental age (eligible if > 12 months).

After qualifying to the study, the screening data will be entered into Biostatistics and Epidemiology Data Analytics Center (BEDAC), secured website. Randomization will then occur. Children will be randomly assigned to one of two intervention options: JASPER + PROMPT versus JASPER only.

JASPER is a naturalistic, developmental, behavioral intervention (NDBI) that focuses on developing social communication and language skills in the context of a play based intervention.

Intervening on oral motor skills may improve speech. In Los Angeles, a fairly common community intervention delivered by certified speech language pathologists (SLP) is Prompts for Restructuring Oral Muscular Phonetic Targets (PROMPT). PROMPT has a growing evidence base among a number of clinical populations with language delays related to oral motor deficits (although not ASD).

1. JASPER only: Child will receive 2, 60 minute sessions per week at UCLA. or
2. JASPER + PROMPT: Child will receive 2, 60 minute sessions per week at Santa Monica's SSLP, Inc.

Recruitment, screening assessments, consents, and treatment will occur in this Santa Monica location for this group. All these procedures will be done by the UCLA staff, except the PROMPT treatment. PROMPT will be done by the SLPs in the Scheflen Speech-Language Pathology, Inc.

All assessments, consent forms, measures, recruitment material will be the same for both conditions.

Interventions will occur for 12 weeks, 3 months. After the 3 months, there will be exit assessments (ELSA Language Sample, PLS-5, ESCS, BOSCC and EEG). There will also be assessment follow up at 3-months post exit, and when the child turns 6 years of age. The following assessments will be done at these time points: ELSA Language Sample, ESCS, BOSCC, PLS-5 at 3 mo-FU and ELSA Language Sample, ESCS, BOSCC, PLS-5 when child turns 6.

ELIGIBILITY:
Inclusion Criteria:

* Children meeting ADOS-2 and ADI-R criteria for ASD
* age 42-66 months
* have had > 3 months of early intervention/preschool (to ensure that children already have been exposed to some community interventions)
* walked prior to 24 months
* use < 20 functional words (i.e., non-echoed, non-scripted). Number of functional spoken words will be totaled in a language sample assessment. The functional word criterion is based on a 2010 NIH workgroup definition of 'minimally verbal' in school-aged children. The same definition may also apply to younger children with limited language.
* stable medication over the past 6 months
* nonverbal mental age of >12 months on the Mullen Scales of Early Learning (visual reception and fine motor subscales).

Exclusion Criteria:

* We will exclude children who are deaf, blind or with cerebral palsy.
* We will not exclude on the basis of known genetic disorder associated with ASD (ex: TSC), but expect few will actually participate, in part due to rarity of these disorders, and because for some there are other trials available at UCLA (ex: TSC).
* We will exclude children in other intervention trials; in other words, we will not double enroll children into intervention trials.

Ages: 42 Months to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in spontaneous socially communicative utterances (SCU) using the Elicitation of Language Samples for Analysis (ELSA). | T1 entry (1st month of study), T2 exit (3 months after entry), T3 3-month Follow Up (6 months after entry), T4 when child turns 6 years of age
  The ELSA is comprised of a series of semi-structured activities including: play-based interactive activities centered around a nature walk (falling leaves; planting an acorn, finding animals; making and eating S'mores); conversational chat and clean up; crafts (art project); games (bean bag toss); and an optional video narration (Pixar short movies, presented to the participant on a tablet).
  The activities are appropriate for the age range of this study (4 to 7 years). The more words the child has, the better the outcome.

SECONDARY OUTCOMES:
Change in number of novel and distinct word root (NDWR), and presence of word combinations at age six based on the ELSA language sample. | T1 entry (1st month of study), T2 exit (3 months after entry), T3 3-month Follow Up (6 months after entry), T4 when child turns 6 years of age
  The ELSA is comprised of a series of semi-structured activities including: play-based interactive activities centered around a nature walk (falling leaves; planting an acorn, finding animals; making and eating S'mores); conversational chat and clean up; crafts (art project); games (bean bag toss); and an optional video narration (Pixar short movies, presented to the participant on a tablet).
  The activities are appropriate for the age range of this study (4 to 7 years). The more words the child has, the better the outcome.
Change in number of novel and distinct word root (NDWR) based on the Preschool Language Scales-5 (PLS-5). | T1 entry (1st month of study), T2 exit (3 months after entry), T3 3-month Follow Up (6 months after entry), T4 when child turns 6 years of age
  A child will be classified verbal if he/she meets the PLS-5 expressive item benchmark for word combinations. Children who do not show word combinations on the Language Sample or PLS-5 will be considered minimally verbal for this analysis.The standard scores for the PLS-5 range from 50 to 150. The higher the score, the better the outcome.
Presence of word combinations at age six based on the Preschool Language Scales-5 (PLS-5) | T1 entry (1st month of study), T2 exit (3 months after entry), T3 3-month Follow Up (6 months after entry), T4 when child turns 6 years of age
  A child will be classified verbal if he/she meets the PLS-5 expressive item benchmark for word combinations. Children who do not show word combinations on the Language Sample or PLS-5 will be considered minimally verbal for this analysis. The standard scores for the PLS-5 range from 50 to 150. The higher the score, the better the outcome.

OTHER OUTCOMES:
Brief Observation of Symptoms of Autism (BOSA) | T1 entry (1st month of study)
  It is a measure that detects the presence or absence of autism symptoms.
Mullen Scales of Early Learning (MSEL) | T1 entry (1st month of study)
  Nonverbal Development Quotients (DQ) (DQ; mental age ÷ chronological age). Raw scores and T-scores are calculated; the higher the number, the better the outcome.
Demographic and Medical Questionnaire | T1 entry (1st month of study)
  Descriptive measure to determine child's eligibility.
Vineland Adaptive Behavior Scale Third Edition (VABS-III) | T1 entry (1st month of study)
  An adaptive behavior assessment. The Adaptive Behavior Composite (ABC) of the VABS-III has a standard score mean of 100 and standard deviation (SD) of 15. Higher scores signifying a better outcome.
Structured Play Assessment-R (SPA) | T1 entry (1st month of study)
  SPA-R is designed to obtain the child's highest levels of spontaneous play acts. The child is presented with 5 different play sets by the experimenter; the entire play interaction last about 15-20 minutes. The child's play behaviors are videotaped and later coded. The variables of interest include the frequency of child initiated functional and symbolic play acts and also the count of different novel types of acts. This measure has shown excellent reliability and validity across a range of studies (Kasari et al., 2006; Sigman & Ruskin, 1999; Sigman & Ungerer, 1984).
Short Sensory Profile (SSP) Questionnaire | T1 entry (1st month of study)
  The Sensory Profile helps you understand a child's sensory processing patterns in everyday situations and profile the sensory system's effect on functional performance for diagnostic and intervention planning. The questionnaire will be filled out by the parent. The questions are scores from 1-5. The higher the score, the better the outcome.
Aberrant Behavior Checklist-2 (ABC-2) | T1 entry (1st month of study)
  The Aberrant Behavior Checklist (ABC) is an informant rating instrument that was empirically derived by principal component analysis (Aman, Singh, Stewart, & Field, 1985a).
Presence of joint attention initiations using the Early Social-Communication Scales | T1 entry (1st month of study), T2 exit (3 months after entry), T3 3-month Follow Up (6 months after entry), T4 when child turns 6 years of age
  In this semi-structured interaction, the child and tester sit facing each other at a table with a set of toys in view but out of reach of the child which are introduced one by one (Mundy, Sigman, Ungerer, & Sherman, 1986; Seibert, Hogan, & Mundy, 1982). The joint attention initiations will then be coded.
Kaufman Speech Praxis Test (KSPT) | T1 entry (1st month of study)
  The KSPT identifies the level of breakdown in a child's ability to speak so that treatment can be established and improvement tracked.
Electroencephalogram (EEG) biomarkers of change with treatment | T1 entry (1st month of study) and T2 exit (3 months after entry)
  The peak alpha frequency will be measured at the beginning of the study and at exit.
Electroencephalogram (EEG) biomarkers of change with treatment | T1 entry (1st month of study) and T2 exit (3 months after entry)
  The frontal gamma power will be measured at the beginning of the study and at exit.
Electroencephalogram (EEG) biomarkers of change with treatment | T1 entry (1st month of study) and T2 exit (3 months after entry)
  The left fronto-temporal alpha will be measured at the beginning of the study and at exit.
Electroencephalogram (EEG) biomarkers of change with treatment | T1 entry (1st month of study) and T2 exit (3 months after entry)
  The gamma coherence will be measured at the beginning of the study and at exit.
Presence of copy-number variations (CNVs) | T1 entry (1st month of study)
  DNA
Polygenetic risk score (PRS) | T1 entry (1st month of study)
  DNA

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Semel Institute, Los Angeles, California
  - UCLA, Los Angeles, California